CLINICAL TRIAL: NCT00988182
Title: The Effect of Whey Protein and Its Hydrolysate on Pre- and Post-Fixed Meal Glycemia and Insulin in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other); Mondelēz International, Inc. (Industry)
Responsible Party: Dr. G. Harvey Anderson, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Kraft_whey protein: study 2
Record Dates: First submitted 2009-09-30; First posted 2009-10-02 (Estimated); Last update posted 2009-10-02 (Estimated); Status verified 2009-10

CONDITIONS: Diabetes Prevention; Obesity Prevention
Keywords: Whey protein; Hydrolysate whey protein; Blood glucose; Insulin
MeSH Terms: conditions — Insulin Resistance | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- whey protein, 5g (Experimental)
  Interventions: Other: dietary intervention
- whey protein, 10g (Experimental)
  Interventions: Other: dietary intervention
- whey protein, 20g (Experimental)
  Interventions: Other: dietary intervention
- whey protein, 40g (Experimental)
  Interventions: Other: dietary intervention
- water control (Experimental)
  Interventions: Other: water control

INTERVENTIONS:
Other: dietary intervention — whey protein
  Arms: whey protein, 10g; whey protein, 20g; whey protein, 40g; whey protein, 5g
Other: water control
  Arms: water control

SUMMARY:
The purpose of this study is to describe relationships among whey protein and its hydrolysate when consumed before a meal on pre- and post-fixed meal satiety, blood glucose and insulin in healthy young adults.

DETAILED DESCRIPTION:
A randomized, cross-over design study was conducted. Whey protein preloads (5-40 g) and hydrolysate whey protein (10 g) were provided in 300 ml water. At 30 min following consumption, subjects were fed a preset pizza meal (12 kcal/kg, experiment 2). Satiety, insulin and blood glucose were measured at baseline and selected intervals pre- and post-meal.

ELIGIBILITY:
Inclusion Criteria:

* normal body weight

Exclusion Criteria:

* breakfast skippers
* smokers
* dieters or individuals with diabetes (fasting blood glucose ≥ 7.0 mmol/L) or other metabolic diseases

Ages: 20 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)

PRIMARY OUTCOMES:
Blood glucose, Insulin, Subjective appetite | 0-170 min

SECONDARY OUTCOMES:
Physical comfort | 0-170 min

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Anderson, Ph.D., Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Department of Nutritional Sciences, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Akhavan T, Luhovyy BL, Brown PH, Cho CE, Anderson GH. Effect of premeal consumption of whey protein and its hydrolysate on food intake and postmeal glycemia and insulin responses in young adults. Am J Clin Nutr. 2010 Apr;91(4):966-75. doi: 10.3945/ajcn.2009.28406. Epub 2010 Feb 17. PMID 20164320